CLINICAL TRIAL: NCT01345123
Title: A Prospective, Randomized Trial to Assess the Impact of Decision Aids and Health Coaching on Health Care Costs, Surgery Rates, and Decision Quality for Individuals At Risk for Musculoskeletal Preference-Sensitive Surgical Decisions
Brief Title: Supporting Decision Making for Musculoskeletal Preference-Sensitive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Dialog (Industry)
Collaborators: Foundation for Informed Medical Decision Making (Other); University of Massachusetts, Boston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDMBKH-HD012011
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-08

CONDITIONS: Knee Pain Chronic; Arthritis (Hip); Arthritis (Knee); Back Pain
MeSH Terms: conditions — Arthritis; Back Pain | interventions — SDM

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Decision Aid with Health Coaching (Experimental)
  Interventions: Behavioral: Provision of condition specific shared decision making (SDM) aids only; Behavioral: Telephonic outreach and support by Health Coach
- Decision Aid only (Experimental)
  Interventions: Behavioral: Provision of condition specific shared decision making (SDM) aids only
- No condition specific support (No Intervention)

INTERVENTIONS:
Behavioral: Provision of condition specific shared decision making (SDM) aids only — Subjects are mailed decision aid digital video discs (DVDs) and pamphlets regarding lumbar back, hip osteoarthritis or knee osteoarthritis.
  Arms: Decision Aid only; Decision Aid with Health Coaching
Behavioral: Telephonic outreach and support by Health Coach — Subjects are direct dial attempted by Health Coaches up to three attempts. If contacted, Health Coaches tailor support around health matters of importance to the subjects and to help individuals become active participants in their treatment plans, and make more informed decisions in consort with their health care providers. The number of total contacts is determined by mutual agreement between the subject and the Health Coach. Health Coaches may provide additional educational materials and resources.
  Arms: Decision Aid with Health Coaching

SUMMARY:
The purpose of this study is to compare condition oriented whole person Health Coaching along with the provision of decision aids to decision aids without condition oriented Health Coaching to neither condition oriented health coaching nor decision aids on medical cost, preference sensitive surgeries and measures of subject knowledge, decision process and decision quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants in two large, commercial Blue Cross and/or Blue Shield branded insurance products with eligibility for Health Dialog services
* Identified by distinct Health Dialog proprietary models for risk of lumbar back, knee or hip surgeries
* Selected by simple randomization for inclusion in an interactive voice response (IVR) administered screening survey
* Participated in an IVR-administered screener survey and responded affirmatively to questions on pain for any one of the three conditions, any current or planned treatment for the conditions, and responded negatively to having had a condition specific surgery within the past six months

Exclusion Criteria:

* People under 18 years of age at time of identification for the IVR filtering survey, approximately 6 weeks prior to the start of the study
* People with invalid phone numbers or invalid mailing addresses based on automated review of those fields
* People for whom Health Dialog has information of a request for no IVR, no Health Coach outreach, or mailings prior to the start of the study
* People with claims based indication of spinal stenosis prior to the start of the study
* People who have been targeted for any IVR outreach within 180 days of the initiation of the IVR filtering survey
* People who have a Health Coach communication record, as documented in the Health Coaching application within 90 days of the start of the study
* Any members of households who have a household member already selected for inclusion in the study
* People for whom there is claims evidence of any one of the targeted surgeries prior the start of the study
* People with no eligibility for services through insurer after the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9925 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Veroff, MPP, Principal Investigator — Health Dialog Services Corporation; Patricia M Gallagher, PHD, Study Director — University of Massachusetts, Boston
Locations (1):
- Health Dialog, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75,795 health plan members recruited via Interactive Voice Response Telephone Call Survey to screen for study eligibility. 30,556 persons completed the screen. 9,925 were study eligible (1. Reported pain in knee, hip, or back; 2. Considering treatment; 3. Had not already had surgery for pain; 4. Not on a 'Do Not Call' list).
Groups:
- Decision Aid With Health Coaching: Study participants receive a digital video disc and booklet (Treatment Choices for Knee Osteoarthritis, Treatment Choices for Hip Osteoarthritis, or Herniated Disc Choosing the right treatment for you) and a call from a nurse health coach.
- Decision Aid Only: Study participants receive a digital video disc and booklet (Treatment Choices for Knee Osteoarthritis, Treatment Choices for Hip Osteoarthritis, or Herniated Disc Choosing the right treatment for you).
- No Condition Specific Support: Study participants do not receive outreach on knee, hip or herniated disc condition.
Period: Overall Study
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Started | 3323 | 3311 | 3291
Completed | 3244 (3323 - 79 study participants who were no longer health plan eligible members (zero eligible months)) | 3226 (3311 - 85 study participants who were no longer health plan eligible members (zero eligible months)) | 3203 (3291 - 88 study participants who were no longer health plan eligible members (zero eligible months))
Not Completed | 79 | 85 | 88
Not completed — participants no longer with health plan | 79 | 85 | 88

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support | Total
Number analyzed (Participants) | 3323 | 3311 | 3291 | 9925
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 2880 | 2922 | 2861 | 8663
  >=65 years | 443 | 388 | 430 | 1261
Age Continuous [Mean (Standard Deviation); unit: years] | 55.94 (10.37) | 56.12 (9.73) | 56.06 (10.14) | 56.04 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1896 | 1888 | 1906 | 5690
  Male | 1427 | 1423 | 1385 | 4235
Region of Enrollment [Number; unit: participants]
  United States | 3323 | 3311 | 3291 | 9925

OUTCOME MEASURES:

1. Primary Outcome: Total Medical Costs Per Member Per Month
Description: total medical cost paid for covered services for the subject for six months after initiation of the study. This total includes all places of service and types of covered services, including inpatient, outpatient and pharmacy.
Time Frame: 6 months
Population: Excluded: Subjects with claim for study-related surgery prior to intervention,claims evidence of symptomatic AIDS, organ transplant, on dialysis, Instituted >= 30days for psych. Subjects with less than 6 months of health plan eligible months. Spinal Stenosis not eligible for study.
Measure: Mean (95% Confidence Interval); unit: Total dollars / member months
Groups:
- Decision Aid Only: Study participants receiving a digital video disc and booklet (Treatment Choices for Knee Osteoarthritis, Treatment Choices for Hip Osteoarthritis, or Herniated Disc Choosing the right treatment for you).
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Number analyzed (Participants) | 2969 | 2942 | 2889
Total dollars / member months | 965.63 [895.66 to 1035.61] | 1000.22 [931.56 to 1068.88] | 965.78 [896.33 to 1035.23]
Statistical Analysis 1: Comparison: Decision Aid With Health Coaching vs No Condition Specific Support; Test type: Superiority or Other; p = 0.9602, ANCOVA; Covariates: age, gender, Charlson Comorbidity Index, prior year total medical costs pmpm; Mean Difference (Net) = 0.00199940, 95% CI 2-sided [-.07658990 to .080588716], Standard Error of Mean .04009180
Statistical Analysis 2: Comparison: Decision Aid Only vs No Condition Specific Support; Test type: Superiority or Other; p = 0.7329, ANCOVA; Mean Difference (Net) = -0.0137170, 95% CI 2-sided [-0.0924947 to 0.06506063], Standard Error of Mean 0.04018791

2. Secondary Outcome: Rate of Targeted Conditions Surgeries
Description: rate of any one claims based instance of lumbar back, hip repair, hip replacement, knee repair, or knee replacement surgery
Time Frame: 6 months
Population: Excluded: Subjects with claim for study-related surgery prior to intervention,claims evidence of symptomatic AIDS, organ transplant, on dialysis, Institutionalized >= 30days for psych. Subjects with less than 6 months of health plan eligible months. Spinal Stenosis not eligible for study.
Measure: Number; unit: percentage of participants
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Number analyzed (Participants) | 2969 | 2942 | 2889
percentage of participants | 5.42 | 6.66 | 6.54
Statistical Analysis 1: Comparison: Decision Aid With Health Coaching vs No Condition Specific Support; Test type: Superiority or Other; p = 0.0511, Regression, Logistic; Covariates: Age, Gender, Charlson Comorbidity index, calculated risk of knee replacement, hip replacement, herniated disc surgery (score 1-99); Odds Ratio (OR) = 0.805, 95% CI [0.647 to 1.001]

3. Secondary Outcome: Concordance
Description: Self-reported consistency of choices with goals and concerns--extent to which the treatment choices subjects make are or are not consistent with the issues they state are priorities including avoiding surgery, reducing pain and regaining function
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Decision Making Process
Description: Self-reported measure of the extent to which subject interactions with providers involve discussions of the pros and cons of treatment options and provide an opportunity for subjects to have input into the decisions.
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Knowledge
Description: Subject self-reported knowledge about the risks and benefits of surgical options and likely outcomes with and without surgical interventions.Knowledge score calculated (score of 0-5, counting number of correct answers) for every respondent who completes at least 3 of the 5 items.
Time Frame: 12 weeks
Population: Decision Quality Survey administered to a random sample (N=2600) of all study participants in the second study wave (N=4208): 1177 survey-eligible respondents, 1124 received a knowledge score.
Measure: Mean (95% Confidence Interval); unit: number of correct answers
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Number analyzed (Participants) | 550 | 354 | 273
number of correct answers | 1.99 [1.8868582 to 2.0942024] | 2.14 [2.0060072 to 2.2805426] | 1.83 [1.6719285 to 1.9894889]
Statistical Analysis 1: Comparison: Decision Aid Only vs No Condition Specific Support; Test type: Superiority or Other; p = 0.0106, ANOVA; Mean Difference (Net) = 0.31257, 95% CI 2-sided [0.06895 to 0.55618]
Statistical Analysis 2: Comparison: Decision Aid With Health Coaching vs No Condition Specific Support; Test type: Superiority or Other; p = 0.0106, ANOVA; Mean Difference (Net) = 0.15982, 95% CI 2-sided [-0.06477 to 0.38441]

6. Secondary Outcome: Decision Conflict
Description: Self-reported measure of the extent to which subjects feel comfortable, supported and confident in choosing one treatment approach over others. Score computed on a scale of 1-3, where 1 = 'No', 2='Yes, somewhat', 3='Yes, completely' (3 indicates less conflict, 1 indicates most conflict) on a 4 item survey question set- asks whether respondents feel sure, have enough support, know and are clear about benefits and risks of treatment options.
Time Frame: 12 weeks
Population: Decision Quality Survey administered to a random sample (N=2600) of all study participants in the second study wave (N=4208): 1177 survey-eligible respondents.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Number analyzed (Participants) | 550 | 354 | 273
units on a scale | 2.2206790 [2.1678803 to 2.2734778] | 2.1876218 [2.1235626 to 2.2516811] | 2.2006866 [2.1260287 to 2.2753446]

7. Secondary Outcome: Decision Satisfaction
Description: Self-reported measure of subject satisfaction with decision as measured retrospectively, including how subjects feel their decision worked out and whether or not they would make the same decision again.
Time Frame: 6 months
Reporting Status: Not Posted

8. Primary Outcome: Total Medical Costs That Can be Impacted Per Member Per Month
Description: total medical cost paid for covered services for the subject for six months after initiation of the study. This total includes all places of service and types of covered services, including inpatient, outpatient and pharmacy.
  Costs that cannot be impacted include: Costs related to Trauma and Accident, Psychiatric/Substance Abuse, Malignant Neoplasm, Maternity and Childbirth excluded
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Total dollars / member months
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Number analyzed (Participants) | 2969 | 2942 | 2889
Total dollars / member months | 679.13 [624.68 to 733.58] | 735.96 [679.55 to 792.37] | 726.88 [665.37 to 788.38]
Statistical Analysis 1: Comparison: Decision Aid With Health Coaching vs No Condition Specific Support; Test type: Superiority or Other; p = 0.8454, ANCOVA; Mean Difference (Net) = -0.0091220, 95% CI 2-sided [-0.1008434 to 0.08259938], Standard Error of Mean 0.04670910
Statistical Analysis 2: Comparison: Decision Aid Only vs No Condition Specific Support; Test type: Superiority or Other; p = 0.6956, ANCOVA; Mean Difference (Net) = -0.0183548, 95% CI 2-sided [-0.1102961 to 0.07358642], Standard Error of Mean 0.04690321

ADVERSE EVENTS:
Arm/Group | Decision Aid With Health Coaching | Decision Aid Only | No Condition Specific Support
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No